CLINICAL TRIAL: NCT05713890
Title: An Integrated and Home-based Motor Rehabilitation Combining Virtual Reality and Action Observation Treatment in People With Multiple Sclerosis: a Clinical and Neuroimaging Study
Brief Title: Home-based Action Observation Treatment With Virtual-reality for Arm Rehabilitation in People With Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Istituto di Neuroscienze Consiglio Nazionale delle Ricerche (Network)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, Professor, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF-2021-12374941
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, single-blinded, parallel study. A total sample size of 60 PwMS is planned, with 30 participants randomly assigned to each of the treatment arms (ratio 1:1) through a computer-generated list managed by a physician external to the study.
Who Masked: Outcomes Assessor
Masking Description: The assessors (neurologists, physiotherapists and neuropsychologists) will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-AOT (Experimental): Home-based Action Observation Treatment with virtual-reality for upper limb rehabilitation
  Interventions: Other: Home-based Action Observation Treatment with virtual-reality for upper limb rehabilitation
- VR-LO (Active Comparator): Home-based landscape observation with virtual-reality for upper limb rehabilitation
  Interventions: Other: Home-based landscape observation with virtual-reality for upper limb rehabilitation

INTERVENTIONS:
Other: Home-based Action Observation Treatment with virtual-reality for upper limb rehabilitation — Observation of a VR scenario depicting multiple repetitions of a specific upper limb motor task belonging to typical activities of daily living, followed by mental imagination of the action observed and then by the execution of the same task, using objects provided in a kit.
  In each session, patients will watch 2 different videos and will perform the two corresponding actions. The time scheduled for observation, imagery and execution of each action will be of 5, 3, and 7 minutes, respectively, so that each session will last about 30 minutes. New actions, chosen from a dataset of 50 stimuli showing progressively increasing levels of difficulty, will be weekly administered on the basis of patient's degree of motor impairment, to involve different manual skills.
  30 minutes sessions, 5 times a week for 3 consecutive weeks (15 sessions in total).
  Arms: VR-AOT
Other: Home-based landscape observation with virtual-reality for upper limb rehabilitation — Observation of virtually explorable landscapes followed by rest with eyes closed without focusing on any thought in particular and then execution of the same actions requested to VR-AOT-group. In each session, patients will explore 2 different landscapes and perform 2 different actions. The time scheduled for observation, rest and action execution will be of 5, 3, and 7 minutes, respectively, so that each session will last about 30 minutes.New actions, chosen from a dataset of 50 stimuli showing progressively increasing levels of difficulty, will be weekly administered on the basis of patient's degree of motor impairment, to involve different manual skills.
  30 minutes sessions, 5 times a week for 3 consecutive weeks (15 sessions in total).
  Arms: VR-LO

SUMMARY:
Action Observation Treatment (AOT) is a rehabilitative strategy which has been proposed as a promising approach to improve motor performance in neurological conditions, including multiple sclerosis (MS).

In this clinical trial, the investigators aim to explore the role of a home-based AOT with virtual reality (VR) in improving upper limb motor function in people with MS (PwMS). The objectives are:

* To compare the effects of home-based VR-AOT versus VR-landscape observation (LO) on upper limb motor performance;
* To measure brain network functional changes (functional plasticity) and structural variations of gray matter (GM) and white matter (WM) (structural plasticity) using advanced magnetic resonance imaging (MRI) techniques following VR-AOT and VR-LO;
* To study the correlations between MRI changes and clinical improvements and the predictors of VR-AOT efficacy.

All participants will undergo treatment sessions for 3 weeks (5 consecutive days/week, total=15 sessions lasting 30 minutes each). Those in the VR-AOT group will observe, imagine and execute two upper limb motor tasks in each session. Those in the VR-LO group will perform the same tasks, but they will observe inanimate landscapes beforehand instead.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years;
* Diagnosis of MS according to 2017 revised McDonald criteria;
* Ability to understand the purpose and risks of the study and provide signed informed consent;
* Ability to remotely perform VR-AOT;
* Right pre-morbid handedness (EHI>50);
* Muscle strength deficit involving the right upper limb (≥1 point decrease of MRC scale);
* Presence of activity limitation of the right hand (need of adaptations, supervision or help by another person for the execution of daily living activities according to items 1-6 of the FIM);
* EDSS score 2.0-7.0 (inclusive);
* Cerebellar functional system score of the EDSS ≤1;
* Baseline 9HPT score >21 seconds and <180 seconds.

Exclusion Criteria:

* MRI contraindications;
* Significant visual deficits not allowing to observe VR stimuli;
* Moderate to severe pain disturbances (VAS≥4);
* Concomitant neuro-psychiatric or systemic diseases (other than MS);
* Clinical relapses or steroid treatment in the past 3 months;
* Modification of symptomatic treatment or botulin toxin injection in the upper limb in the past 3 months;
* Stable disease-modifying treatment for MS for ≤6 months;
* Rehabilitation treatment in the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in right hand Nine-hole peg test (9HPT) | Baseline, after 3 weeks of training and after a 3-month follow-up
  Time required to complete the 9HPT, a measure of hand dexterity, with the right hand (average of two tests).

SECONDARY OUTCOMES:
Change in left hand Nine-hole peg test (9HPT) | Baseline, after 3 weeks of training and after a 3-month follow-up
  Time required to complete the 9HPT, a measure of hand dexterity, with the left hand (average of two tests).
Change in hand grip strength | Baseline, after 3 weeks of training and after a 3-month follow-up
  Hand grip strength measured with the Jamar handheld dynamometer. Measured for left and right hand separately.
Change in finger tapping frequency | Baseline, after 3 weeks of training and after a 3-month follow-up
  Number of taps performed with the index finger in 30 seconds (average of two trials). Measured for left and right hand separately.
Change in Medical Research Council (MRC) scale | Baseline, after 3 weeks of training and after a 3-month follow-up
  Segmental upper limb strength measured using the MRC scale. Scores on this scale range from 0 (no visible contraction) to 5 (normal strength). Measured for left and right upper limb separately.
Change in Modified Ashworth Scale (MAS) | Baseline, after 3 weeks of training and after a 3-month follow-up
  Upper limb spasticity (shoulder adductors, elbow flexors, wrist flexors and pronators) measured using the MAS. Scores in this scale range from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension). Measured for left and right upper limb separately.
Change in items 1-6 of the Functional Independence Measure (FIM) | Baseline, after 3 weeks of training and after a 3-month follow-up
  Autonomy in upper limb-related activities of daily living measured with items 1-6 of the FIM. Each item's score ranges from 1 (total assistance needed) to 7 (complete independence).
Change in Expanded Disability Status Scale (EDSS) | Baseline, after 3 weeks of training and after a 3-month follow-up
  Multiple sclerosis-related global disability and functional systems subscores. Scores in this scale range from 0 (normal neurological function) to 10 (death due to multiple sclerosis).
Change in Paced Auditory Serial Addition Test (PASAT) | Baseline, after 3 weeks of training and after a 3-month follow-up
  A cognitive task that measures sustained attention and working memory. The scores of this test, ranging from 0 to 60, are corrected for age, sex and years of education. Higher scores reflect a better performance in the test.
Change in Symbol-Digit Modalities Test (SDMT) | Baseline, after 3 weeks of training and after a 3-month follow-up
  A cognitive task that measures information processing speed. The scores of this test, ranging from 0 to 110, are corrected for age, sex and years of education. Higher scores reflect a better performance in the test.
Change in Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline, after 3 weeks of training and after a 3-month follow-up
  An instrument that rates the severity of depressive symptoms. It is administered by a clinician through an interview. It is composed by 10 items, each with a score ranging from 0 to 6. The overall score ranges from 0 to 60, with higher scores reflecting greater severity of depressive symptoms.
Change in Modified Fatigue Impact Scale (MFIS) | Baseline, after 3 weeks of training and after a 3-month follow-up
  A 21-item scale where patients rate their perceived feeling of fatigue in three subscales (physical, cognitive and psychosocial). The total score of this scale ranges from 0 to 84, with higher scores reflecting more impact of fatigue in everyday life.
Change in Arm Function in Multiple Sclerosis Questionnaire (AMSQ) | Baseline, after 3 weeks of training and after a 3-month follow-up
  A self-reported measure of upper limb function containing 31 items. The score of this scale ranges from 31 to 186, with higher scores indicating more limitation in hand and arm function.
Change in Multiple Sclerosis Quality of Life-54 (MSQOL-54) | Baseline, after 3 weeks of training and after a 3-month follow-up
  A health-related measure of quality of life in people with MS. It contains 54 items grouped in 12 subscales. Two summary scores can be extracted from this scale: the physical health and mental health composite scores. These scores can be derived from a weighted combination of scale scores (scale scores range from 0 to 100 and a higher scale score indicates better quality of life).
Change in global brain volume | Baseline and after 3 weeks of training
  Normalized volumes of the brain, GM and WM will be extracted from 3D T1 MRI sequences.
Changes in regional gray matter volumes | Baseline and after 3 weeks of training
  Tensor-based morphometry (TBM) will be used to map and compare longitudinal changes of regional GM volumes between groups
Changes in white matter microstructural architecture | Baseline and after 3 weeks of training
  Tract-based spatial statistics (TBSS) will be used to map training-related changes of WM architecture.
Changes in resting state functional connectivity | Baseline and after 3 weeks of training
  Independent Component Analysis will be used to decompose resting state functional MRI data into spatially independent maps and time courses, and to select the main sensory and motor functional networks of interest, as well as the Mirror Neuron System network.
Changes in brain activation during an object manipulation task | Baseline and after 3 weeks of training
  Statistical Parametric Mapping (SPM) 12 will be applied to functional MRI sequences acquired during the object manipulation task to evaluate the modifications of functional activations during this task.

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Rocca, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The dataset including all the data obtained from this study will be available from the Principal Investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The dataset including all the data obtained from this study will be available 6 months after the publication of the results.
Access Criteria: The dataset including all the data obtained from this study will be available from the Principal Investigator upon reasonable request.

REFERENCES:
- [Background] Rocca MA, Tortorella P, Ceccarelli A, Falini A, Tango D, Scotti G, Comi G, Filippi M. The "mirror-neuron system" in MS: A 3 tesla fMRI study. Neurology. 2008 Jan 22;70(4):255-62. doi: 10.1212/01.wnl.0000284667.29375.7e. Epub 2007 Dec 12. PMID 18077798
- [Background] Rocca MA, Meani A, Fumagalli S, Pagani E, Gatti R, Martinelli-Boneschi F, Esposito F, Preziosa P, Cordani C, Comi G, Filippi M. Functional and structural plasticity following action observation training in multiple sclerosis. Mult Scler. 2019 Oct;25(11):1472-1487. doi: 10.1177/1352458518792771. Epub 2018 Aug 7. PMID 30084706
- [Background] Rizzolatti G, Fabbri-Destro M, Nuara A, Gatti R, Avanzini P. The role of mirror mechanism in the recovery, maintenance, and acquisition of motor abilities. Neurosci Biobehav Rev. 2021 Aug;127:404-423. doi: 10.1016/j.neubiorev.2021.04.024. Epub 2021 Apr 25. PMID 33910057
- [Background] Nuara A, Avanzini P, Rizzolatti G, Fabbri-Destro M. Efficacy of a home-based platform for child-to-child interaction on hand motor function in unilateral cerebral palsy. Dev Med Child Neurol. 2019 Nov;61(11):1314-1322. doi: 10.1111/dmcn.14262. Epub 2019 May 21. PMID 31115046
- [Background] De Marco D, Scalona E, Bazzini MC, Nuara A, Taglione E, Lopomo NF, Rizzolatti G, Fabbri-Destro M, Avanzini P. Observation of others' actions during limb immobilization prevents the subsequent decay of motor performance. Proc Natl Acad Sci U S A. 2021 Nov 23;118(47):e2025979118. doi: 10.1073/pnas.2025979118. PMID 34782480
- [Background] Jonsdottir J, Perini G, Ascolese A, Bowman T, Montesano A, Lawo M, Bertoni R. Unilateral arm rehabilitation for persons with multiple sclerosis using serious games in a virtual reality approach: Bilateral treatment effect? Mult Scler Relat Disord. 2019 Oct;35:76-82. doi: 10.1016/j.msard.2019.07.010. Epub 2019 Jul 20. PMID 31352180